CLINICAL TRIAL: NCT04713163
Title: Prospective Evaluation of COVID-19 Vaccine Induced Immunity
Brief Title: COVID-19 Vaccine Induced Immunity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); Cadham Provincial Lab (Unknown)
Responsible Party: Principal Investigator, Lyle Mckinnon, Assistant Professor, University of Manitoba
Other Study IDs: B2021:008
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Health care or laboratory-based workers: Healthy individuals about to receive any approved COVID-19 vaccine
  Interventions: Drug: covid19 vaccine
- Outpatients: Outpatients about to receive any approved COVID-19 vaccine
  Interventions: Drug: covid19 vaccine

INTERVENTIONS:
Drug: covid19 vaccine — Vaccine
  Other Names: moderna or Pfizer mRNA vaccines, or any other vaccine for Covid19 that becomes approved in Canada

SUMMARY:
This study aims to address the following three objectives:

1. Longitudinal evaluation of the development of CMI responses in response to SARS-CoV-2 Vaccine: T cells isolated from the blood of COVID-19 vaccine recipients will be evaluated for their functionality in response to vaccine antigens. The temporal and functional properties of CMI responses will be correlated with the humoral or antibody responsiveness. CMI responses will be measured in vaccine recipients prior to vaccination to determine whether the presence or functionality of pre-existing responses to common cold coronaviruses (CCCs) or previous SARS-CoV-2 infections affect the development of CMI responses to the COVID-19 vaccine.
2. Identification of cellular and soluble factors that influence vaccine responsiveness:

   While it is known that poor clinical outcomes in COVID-19 patients are strongly associated with markers of systemic inflammation, the influence these systemic markers will have on COVID-19 vaccine responsiveness is not clear. Using systems biology approaches, the investigators will perform comprehensive profiling of cellular immune subsets, inflammatory signatures to identify determinants influencing the development of CMI responses to vaccine.
3. Examine variability of immune and viral genes and their relationship to vaccine induced immune responses: Human leukocyte antigen (HLA), T cell receptor (TCR) and B cell receptor (BCR) proteins are highly genetically diverse and critical to development of protective immunity. The investigators will perform HLA sequencing on whole blood-derived DNA samples and TCR and BCR sequencing on sorted, SARS-CoV2 vaccine antigen-specific T cells and B cells, respectively, to assess how different sequence combinations impact the CMI responses to vaccine.

ELIGIBILITY:
Inclusion Criteria:

* all individuals eligible to receive one of the approved SARS-CoV-2/COVID-19 vaccines.

Exclusion Criteria:

* individuals under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers eligible to receive Covid-19 vaccines
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Nasal T cell responses | Change from Baseline to 12 days post second vaccine dose
  Phenotype of CD4 and CD8+ T cells measured by nasal swabs
Systemic T cell responses | Change from Baseline to 12 days post second vaccine dose
  Cytokine responsiveness to SARS-CoV-2-specific CD4 and CD8+ T cells in blood
Systemic and nasal antibody responses | Change from Baseline to 12 days post second vaccine dose
  IgA and IgG responses to SARS-CoV-2

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT04713163/Prot_SAP_000.pdf